CLINICAL TRIAL: NCT05344235
Title: Observational Study on Extreme Hypofractionation for Localized Prostate Cancer
Acronym: OBELIX PCa
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S66399
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer; Radiotherapy; SBRT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: SBRT — stereotactic radiotherapy of the primary prostate

SUMMARY:
Radiotherapy (RT) is an established treatment option for localized prostate cancer (PCa), with cure rates similar to those of radical prostatectomy. In the last decade, conventionally fractionated RT (1.8-2.0 Gy per fraction to 78-80 Gy) has been replaced by moderately hypofractionated RT (2.3-3.65 Gy per fraction to 56-70 Gy). The rationale behind this change is the scientific level 1 evidence that a higher dose per fraction may improve the cost-benefit of RT due to the specific radiobiology of PCa (a lower alpha/beta than that of adjacent healthy tissues). Additionally, there is a practical advantage both for patients and the radiation department due to a reduced number of fractions.

More recently, extreme hypofractionation or stereotactic body radiotherapy (SBRT) (7-9.5 Gy per fraction to 36-43 Gy in 4-7 fractions) has been introduced as RT modality, and proved to be an effective and safe treatment option for patients with low and intermediate clinically-localized PCa, with similar incidence of late toxicity and 5-year disease free survival outcomes when compared to hypofractionated and conventional radiotherapy regimens. International guidelines endorse extreme hypofractionated SBRT as routine treatment option for low and intermediate risk PCa patients. For high-risk prostate cancer, preliminary results of ongoing prospective studies are promising, but these data are not yet mature enough to recommend extreme hypofractionated SBRT in high-risk prostate cancer. Upon this, ongoing prospective trials handle strict eligibility criteria hereby selecting patients with few comorbidities. This may not necessarily fully reflect the real life patient population. Indeed, patients with a large prostate size, a history of transurethral resection of the prostate (TURP), or 'significant' urinary baseline symptoms may be at risk for experiencing increased toxicity. Based on this concern, these patients were excluded from ongoing clinical trials. However, whether these patients will really develop more toxicity, is a theoretical concern, not yet based on clinical evidence. It is our hypothesis that using modern radiotherapy such as volumetric arc therapy (VMAT) and image-guided radiotherapy (IGRT) - both standard technologies at the Radiation-Oncology department in Leuven University Hospitals - extreme hypofractionated SBRT can be successfully implemented in the treatment of intermediate risk and a select group of high-risk PCa patients and/or patients with pre-existing urinary morbidity.

ELIGIBILITY:
Inclusion Criteria:

* men ≥ 18 years
* histologically confirmed clinically localized adenocarcinoma of the prostate
* intermediate- or high-risk PCa, defined as

OR at least one of the following criteria:

* clinical stage: cT2a-c, cT3a or cT3b (AJCC 7th edition)
* Gleason Score ≥ 7 (ISUP grade group 2 or higher)

OR at least two of the following criteria:

* clinical stage: cT1c (AJCC 7th edition)
* Gleason Score ≥ 7 (ISUP grade group 2 or higher)
* calculated risk for lymph node involvement (Roach formula) <35%.
* no evidence of disease spread beyond the prostate and/or seminal vesicles
* imaging with mpMRI of the prostate and pelvis (compliant with the PIRADS v2.1 guidelines) within 90 days prior to registration, or required to be performed after registration to the trial
* ability to understand, and willingness to sign, the written informed consent
* willingness to comply with scheduled visits, treatment, and other procedures

Exclusion Criteria:

* prior pelvic irradiation (external beam radiotherapy or brachytherapy)
* previous radical prostatectomy, cryosurgery, or HIFU for prostate cancer
* previous or concurrent cytotoxic chemotherapy for prostate cancer
* patients with neuroendocrine or small cell carcinoma of the prostate
* clinical stage cT4 (invasion of adjacent organ like bladder or rectum, visualized on mpMRI and/or ultrasound and endoscopy) (AJCC 7th edition)
* significant urinary obstruction of other voiding symptoms (IPSS > 18) is allowed, however should be discussed with the principal investigator and left to the discretion of the treating physician
* high risk of lymph node involvement, as calculated with the Roach formula ≥ 35% (https://www.evidencio.com/models/show/1144) Of note, in case of ambiguity of regional lymph node involvement on CT or MRI findings (when Roach formula is < 35%, and all other eligibility criteria are met), dedicated imaging with PSMA PET-CT or extended pelvic lymph node dissection must be obtained to rule out lymph node involvement
* evidence of distant metastases (based on CT scan, MRI of the pelvis, bone scan within 90 days prior to registration; if the bone scan is suspicious but not unequivocal, dedicated X-ray and/or MRI must be obtained to rule out metastasis)
* contraindications to MRI according to the Radiology Department guidelines (metal implants, noncompatible cardiac device, deep brain stimulators, cochlear implants, metallic foreign body in the eye or aneurysm clips in the brain, severe claustrophobia).
* World Health Organization (WHO) performance score > 2
* patients with severe inflammatory bowel disease rendering radiotherapy impossible (active Crohn's Disease or Ulcerative Colitis), or patients known with ataxia telangiectasia
* implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion
* prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease-free for a minimum of 5 years.

(carcinoma in situ of the bladder or oral cavity is permissible)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — only males can be included in the trial
Study Population: localized intermediate or high risk prostate cancer (Roach formule < 35%) (cT1-3a/b cN0 M0)
Sampling Method: Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
acute toxicity | toxicity occurring within 90 days after the first SBRT session
  acute gastrointestinal (GI) and genitourinary (GU) Common Terminology Criteria for Adverse Events version 5.0 (CTCAE 5.0)

SECONDARY OUTCOMES:
late toxicity | 90 days to 5 years after the last radiation treatment
  late GI and GU CTCAE v5.0
impact on quality if of life | until month 60
  questionnaires EORTC QLQ-C30, EORTC PR25
(Biochemical and Clinical) Relapse-free survival | until month 60
  Biochemical disease-free survival will be assessed using the Phoenix consensus definition (time frame = 5 years). Clinical relapse-free survival will be defined by the occurrence of any clinical relapse (local, nodal or distant) captured on state-of-the-art imaging (PSMA PET-CT) and triggered by biochemical recurrence and/or occurrence of disease-related symptoms, or in case of accidental findings on imaging performed for other indications (Kaplan Meier statistics).
Dose-volume parameters | until month 60
  dose to the organs at risk (Gray, unit)

CONTACTS AND LOCATIONS:
Overall Officials: Gert De Meerleer, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
no sharing of IPD due to GDPR